CLINICAL TRIAL: NCT07265128
Title: Effect of Remimazolam on Delirium After Cardiac Surgery: Randomized Controlled Trial With Midazolam
Brief Title: Remimazolam vs Midazolam to Reduce Delirium in Adults ≥65 Undergoing CPB Valve Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2024-0976
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Delirium; Critical Illness; Aged; Cardiopulmonary Bypass; Benzodiazepines
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Midazolam; Control Groups; remimazolam

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group comparison of remimazolam versus midazolam for anesthetic induction in adults over 65yrs undergoing cardiopulmonary bypass valve surgery to evaluate postoperative delirium.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design in which participants, care providers, investigators, and outcome assessors are unaware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam group (Active Comparator): Patients allocated to receive midazolam during anesthetic induction and rewarming period of cardiopulmonary bypass.
  Interventions: Drug: Midazolam
- Remimazolam group (Experimental): Patients allocated to receive remimazolam during anesthetic induction and rewarming period of cardiopulmonary bypass.
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Midazolam — Participants receive intravenous midazolam 0.05 mg/kg for anesthetic induction and an additional dose (0.065 mg/kg) administered via the cardiopulmonary bypass circuit during rewarming, with all other anesthetic management identical to the experimental arm.
  Other Names: Control group
  Arms: Midazolam group
Drug: Remimazolam — Participants receive intravenous remimazolam 0.2 mg/kg for anesthetic induction and an additional dose (0.26 mg/kg) administered via the cardiopulmonary bypass circuit during rewarming, together with standard cardiac anesthesia care.
  Other Names: Byfavo group
  Arms: Remimazolam group

SUMMARY:
"Postoperative delirium is a common and serious complication following cardiac surgery, particularly among older adults who require intensive care. Its incidence is reported to range between 20% and 70% after cardiopulmonary bypass (CPB), and has been associated with prolonged hospitalization, increased medical costs, higher morbidity and mortality, and long-term cognitive decline. Benzodiazepines are frequently used during anesthetic induction in cardiac surgery due to favorable hemodynamic stability, although multiple clinical guidelines have recommended limitation of benzodiazepine exposure because of concerns for delirium. However, robust clinical evidence in cardiac surgery remains limited.

Midazolam is currently the most commonly administered benzodiazepine in this setting, though metabolism through hepatic pathways and accumulation of active metabolites may increase the risk of postoperative delirium, especially in older patients and those with organ dysfunction. Remimazolam, a recently approved benzodiazepine, undergoes rapid hydrolysis by plasma esterases and demonstrates predictable pharmacokinetic properties with a markedly shorter context-sensitive half-time compared to midazolam. These pharmacologic features suggest a potentially reduced impact on postoperative delirium risk. Despite this rationale, no randomized controlled trial has evaluated the effect of remimazolam versus midazolam on delirium after CPB-assisted valve surgery.

This randomized double-blind controlled trial aims to determine whether remimazolam reduces the incidence of postoperative delirium compared with midazolam in patients aged ≥65 years undergoing valve surgery with CPB. Eligible participants will be randomized in a 1:1 ratio to receive either remimazolam or midazolam for anesthetic induction according to a computer-generated allocation sequence. All other anesthetic management will follow standardized institutional protocols, including depth of anesthesia monitoring. Delirium assessment will be performed three times daily in the intensive care unit using Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or Intensive Care Delirium Screening Checklist (ICDSC) and twice daily on the ward using 3-Minute Diagnostic Interview for CAM (3D-CAM) for four postoperative days.

The primary endpoint is the incidence of delirium within four postoperative days. Key secondary outcomes include in-hospital or 30-day mortality and a composite of major postoperative complications. A total of 300 patients (150 per group) will be enrolled to provide 90% statistical power to detect the hypothesized difference in delirium risk between groups, accounting for a 10% dropout rate. Findings from this study are expected to provide high-quality evidence regarding the comparative impact of remimazolam and midazolam on postoperative delirium and may inform anesthetic strategy selection in high-risk cardiac surgical populations."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older undergoing heart valve surgery involving cardiopulmonary bypass.

Exclusion Criteria:

* Emergency surgery, Surgery involving total arch replacement, History of remimazolam anaphylaxis, History of major neurocognitive disorder, Alcohol or substance dependence/abuse, Major depressive disorder, Schizophrenia, Participation in other clinical studies that may affect outcomes, Inability to provide informed consent due to illiteracy, foreign language barrier, or cognitive impairment.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium within 4 days after surgery | From the day of surgery (POD 0) to postoperative day 4
  Occurrence of delirium assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU), Intensive Care Delirium Screening Checklist (ICDSC), or 3-Minute Diagnostic Interview for CAM (3D-CAM) during the first 4 postoperative days.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided